CLINICAL TRIAL: NCT01827787
Title: A Phase 2 Study of Eribulin in Patients With HER2-Negative, Metastatic Breast Cancer: Evaluation of Efficacy, Toxicity and Patient-Reported Outcomes
Brief Title: Eribulin in HER2 Negative Metastatic BrCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-077
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Intervention Model Description: This is not a randomized trial rather participants are enrolled based on disease histology. Participants in each arm receive the same treatment regimen.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: HR+/HER2- (Experimental): Eribulin: 1.4 mg/m2 administered intravenously over 2-5 minutes on days 1 and 8 of each 21 day cycle
  Participants remained on single agent eribulin until disease progression or withdrawal for other reasons.
  Interventions: Drug: Eribulin
- Cohort 2: TNBC (Experimental): Eribulin: 1.4 mg/m2 administered intravenously over 2-5 minutes on days 1 and 8 of each 21 day cycle
  Participants remained on single agent eribulin until disease progression or withdrawal for other reasons.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin
  Other Names: E7389; Halaven; ER-086526; NSC-707389

SUMMARY:
Improvements in outcomes with metastatic breast cancer (MBC) have been observed in the last 30 years, however, overall prognosis remains poor with median survival of 2 to 3 years. Long term complete responses are observed only for a minority of MBC patients (2-5%) and MBC remains an incurable disease for most patients. Eribulin is a chemotherapy approved by the US FDA in November of 2010 to treat patients with MBC who have received at least two prior chemotherapy regimens. In this research study, the investigators are looking to see how well eribulin helps participants with MBC in an earlier-line setting. Eribulin works by interfering with cancer cell division, growth and spread.

DETAILED DESCRIPTION:
Based on positive results in heavily pre-treated MBC patients, eribulin is being studied as first-line or second-line chemotherapy treatment. This is a non-randomized, open label study with participants enrolled in one of two cohorts: Cohort 1. Hormone receptor (HR)-positive/human epidermal growth factor receptor 2 (HER2)-negative (HR+/HER2-) or Cohort 2: Triple negative breast cancer (TNBC) meaning HR-negative/HER2-negative (HR-/HER2-). HR- means progesterone receptor-negative (PR-) and estrogen receptor-negative (ER-). Beyond efficacy as measured primarily by response to treatment, investigators will evaluate safety, tolerability and quality of life. In particular, it is hypothesized that eribulin may have lower rates of neuropathy, a common side effect of many of the major chemotherapeutics with activity in MBC. The investigators will study the effect eribulin has on the nerves through regular questionnaires that ask about any nerve-related symptoms. The investigators also plan to send blood samples to explore if gene markers may indicate increased sensitivity to the nerve effects of eribulin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven invasive breast cancer, locally recurrent or metastatic, with at least one measureable lesion according to RECIST v1.1
* Hormone receptor positive or hormone receptor negative HER2-negative disease
* Up to one prior line of chemotherapy for advanced disease is allowed (discontinued at least 14 days prior to initiation of protocol therapy)
* Prior bevacizumab in the neo/adjuvant or metastatic setting is acceptable
* No limit on prior lines of endocrine therapy, but must be discontinued at least 7 days prior to initiation of protocol therapy
* Must have completed any prior radiotherapy at least 2 weeks prior to initiation of protocol therapy
* Must have recovered from reversible effects of prior therapies to no more than grade 1 toxicity, with the exception of alopecia
* Agree to use adequate contraception for the duration of study participation

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior treatment with eribulin
* Prior malignancy other than carcinoma in situ of the cervix or nonmelanoma skin cancer unless diagnosed and definitively treated at least 3 years before enrollment in this study
* Clinically significant cardiovascular impairment
* Active brain metastases or unevaluated neurologic symptoms suggestive of brain metastases
* Pulmonary dysfunction requiring the use of oxygen
* Prior organ allograft requiring immunosuppression
* HIV positive on combination antiretroviral therapy
* Pre-existing grade 3 or 4 neuropathy
* Hypersensitivity to halichondrin B or halichondrin B chemical derivative
* Uncontrolled intercurrent illness
* Inability to read in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Eastern Maine Medical Center, Bangor, Maine
  - Dana-Farber Cancer Institute at Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - DF/BWCC at Milford Regional Cancer Center, Milford, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filho OM, Giobbie-Hurder A, Lin NU, Faggen M, Come S, Openshaw T, Constantine M, Walsh J, Freedman RA, Schneider B, Burstein HJ, Mayer EL. A dynamic portrait of adverse events for breast cancer patients: results from a phase II clinical trial of eribulin in advanced HER2-negative breast cancer. Breast Cancer Res Treat. 2021 Jan;185(1):135-144. doi: 10.1007/s10549-020-05928-4. Epub 2020 Oct 6. PMID 33025482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between May 2013 and March 2016.
Period: Overall Study
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Started | 45 | 38
Completed | 45 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC | Total
Number analyzed (Participants) | 45 | 38 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 33 | 68
  >=65 years | 10 | 5 | 15
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 87] | 53 [38 to 76] | 56 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 35 | 76
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 42 | 34 | 76
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 45 | 38 | 83
Eastern Cooperative Oncology Group Performance Score (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours
  Participants
    ECOG PS0 | 33 | 26 | 59
    ECOG PS1 | 11 | 12 | 23
    ECOG PS2 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 9 weeks on treatment; Maximum treatment duration was 38 cycles/26 months (Cohort 1) and 17 cycles/12 months (Cohort 2)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Number analyzed (Participants) | 45 | 38
percentage of participants | 35.6 [24 to 49] | 13.2 [5 to 26]
Statistical Analysis 1: Comparison: Cohort 1: HR+/HER2-; Using a one sample binomial design, with 45 patients there was 90% power to detect a null hypothesis 30% overall response rate (historical control) versus an alternative hypothesis of 53% overall response rate assuming a two-sided 10% alpha. Of note, cohort 2: TNBC did not fully accrue 45 patients so a testing was not done; Test type: Superiority; p = 0.42, Fisher Exact

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD are censored at date of last disease assessment. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum longest diameter (LD), taking as reference the smallest sum on study with at least 5 mm absolute increase or the appearance of one or more new lesions. For non-target lesions, PD is appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 9 weeks on and off treatment; Median (maximum) PFS follow-up was 12.6 (27.1) months in Cohort 1 and 12.4 (14.3) months in Cohort 2.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Mean (90% Confidence Interval); unit: months
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Number analyzed (Participants) | 45 | 38
months | 6.2 [5.9 to 8.7] | 4.0 [3.5 to 4.8]

3. Secondary Outcome: Time to First Response (TTR)
Description: TTR is defined as the time from first dose of study treatment until the earliest date that complete response (CR) or partial response (PR) based on RECIST 1.1 criteria is objectively documented. Non-CR, non-PR participants are censored at date of last disease assessment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response requires 4 week or later confirmation and assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Number analyzed (Participants) | 45 | 38
months | 10.6 [1.7 to 14.9] | NA [1.9 to 4.3] — Median was not reached.

4. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR is defined as the that response criteria for CR or PR (whichever is recorded first) are first met until the date that PD or death from any cause is first objectively documented. Participants who do not have PD will be censored on date of last disease assessment.
Time Frame: Disease was evaluated radiologically at baseline and every 9 weeks on and off treatment; Median (maximum) DOR follow-up was 12.6 (27.1) months in Cohort 1 and 12.4 (14.3) months in Cohort 2.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Number analyzed (Participants) | 45 | 38
months | 6.5 [1.8 to 12.3] | 1.9 [1.3 to 4.1]

5. Secondary Outcome: Percentage of Participants With Grade 1-3 Treatment-Related Peripheral Sensory Neuropathy
Description: The percentage of treated participants experiencing grade 1-3 peripheral sensory neuropathy with treatment attribution of possible, probable or definite based on Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) as reported on case report forms.
Time Frame: Adverse events were assessed every cycle throughout treatment. Maximum treatment duration was 38 cycles/26 months (Cohort 1) and 17 cycles/12 months (Cohort 2)
Population: The analysis dataset is comprised of all treated participants. Per protocol, the cohorts were combined for this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Combined Cohort 1: HR+/HER2- and Cohort 2: TNBC: Eribulin: 1.4 mg/m2 administered intravenously over 2-5 minutes on days 1 and 8 of each 21 day cycle
  Participants remained on single agent eribulin until disease progression or withdrawal for other reasons.
Arm/Group | Combined Cohort 1: HR+/HER2- and Cohort 2: TNBC
Number analyzed (Participants) | 83
percentage of participants | 36.1 [27.4 to 45.7]

6. Secondary Outcome: Percentage of Participants With Grade 1-3 Treatment-Related Peripheral Motor Neuropathy
Description: TThe percentage of treated participants experiencing grade 1-3 peripheral motor neuropathy with treatment attribution of possible, probable or definite based on Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) as reported on case report forms.
Time Frame: as for outcome 5
Population: The analysis dataset is comprised of all treated participants.Per protocol, the cohorts were combined for this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Cohort 1: HR+/HER2- and Cohort 2: TNBC
Number analyzed (Participants) | 83
percentage of participants | 22.9 [15.5 to 31.7]

7. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast Cancer Subscale (FACT-BCS) Change Score From Baseline
Description: The FACT-BCS is a validated, self-administered questionnaire which captures quality of life (QOL) concerns specific to breast cancer patients. (Brady MJ, et al. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. JCO 1997; 15:974-86). The FACT-BCS has 9-items scored on a 5-point Likert scale (Not at all, A little bit, Somewhat, Quite a bit, Very much) with a maximum score of 36. A higher score indicates better QOL. A minimal clinically important difference is 3-5 points.
Time Frame: Assessed at baseline and on treatment day 1 of cycles 2, 3, 5, 7, 9 and 11
Population: The analysis dataset is comprised of all participants who completed both QOL assessments required to calculate change from baseline. Per protocol, the cohorts were combined for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combined Group (Hormone Receptor Positive and Triple Negative): Eribulin Monotherapy
  Eribulin: Intravenously on Day 1 and 8 of each cycle
Arm/Group | Combined Group (Hormone Receptor Positive and Triple Negative)
Number analyzed (Participants) | 83
units on a scale
  Cycle 2 Change from Baseline: number analyzed (Participants) | 43
  Cycle 2 Change from Baseline | 1.0 (4.6)
  Cycle 3 Change from Baseline: number analyzed (Participants) | 40
  Cycle 3 Change from Baseline | 0.6 (5.1)
  Cycle 5 Change from Baseline: number analyzed (Participants) | 26
  Cycle 5 Change from Baseline | 0.1 (4.4)
  Cycle 7 Change from Baseline: number analyzed (Participants) | 18
  Cycle 7 Change from Baseline | 0.6 (3.2)
  Cycle 9 Change from Baseline: number analyzed (Participants) | 13
  Cycle 9 Change from Baseline | 1.8 (5.0)
  Cycle 11 Change from Baseline: number analyzed (Participants) | 9
  Cycle 11 Change from Baseline | 1.1 (2.9)

8. Secondary Outcome: Functional Assessment of Cancer Therapy-Neurotoxicity Subscale (FACT-Ntx) Change Score From Baseline
Description: The FACT-Ntx is a validated, self-administered questionnaire which captures quality of life (QOL) concerns specific to patients suffering from neurotoxicity. (Calhoun EA, et al. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer 2003; 13:741-8). The FACT-Ntx has 11-items scored on a 5-point Likert scale (Not at all, A little bit, Somewhat, Quite a bit, Very much) with a maximum score of 44. A higher score indicates better QOL. A minimal clinically important difference is 3-5 points.
Time Frame: Assessed at baseline and on treatment day 1 of cycles 2, 3, 5, 7, 9 and 11
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combine Cohort 1: HR+/HER2- and Cohort 2: TNBC: Eribulin: 1.4 mg/m2 administered intravenously over 2-5 minutes on days 1 and 8 of each 21 day cycle
  Participants remained on single agent eribulin until disease progression or withdrawal for other reasons.
Arm/Group | Combine Cohort 1: HR+/HER2- and Cohort 2: TNBC
Number analyzed (Participants) | 83
units on a scale
  Cycle 2 Change from Baseline | -0.1 (3.0)
  Cycle 3 Change from Baseline | -0.3 (4.7)
  Cycle 5 Change from Baseline | -1.6 (5.5)
  Cycle 7 Change from Baseline | -4.5 (6.4)
  Cycle 9 Change from Baseline | -1.8 (5.9)
  Cycle 11 Change from Baseline | -1.6 (4.7)

9. Post Hoc Outcome: Overall Survival
Description: OS based on Kaplan-Meier is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Overall median survival follow-up was 5.9 months including a maximum of 27 months for Cohort 1 and 15 months for Cohort 2.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
Number analyzed (Participants) | 45 | 38
months | 20 [20 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 90% CI. | 11.3 [9.1 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 90% CI.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed every cycle on treatment. Maximum treatment duration was 38 cycles/26 months (Cohort 1) and 17 cycles/12 months (Cohort 2).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | Cohort 1: HR+/HER2- | Cohort 2: TNBC
All-Cause Mortality (participants affected / at risk) | 4/45 | 9/38
Serious Adverse Events (participants affected / at risk) | 22/45 | 13/38
Other Adverse Events (participants affected / at risk) | 45/45 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: HR+/HER2- (N=45) | Cohort 2: TNBC (N=38)
Alkaline phosphatase increased (Investigations) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Lip infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 16 | 4
Peripheral motor neuropathy (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Thromboembolic event (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
White blood cell decreased (Investigations) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: HR+/HER2- (N=45) | Cohort 2: TNBC (N=38)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Alanine aminotransferase increased (Investigations) | 8 | 4
Alkaline phosphatase increased (Investigations) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 15
Anemia (Blood and lymphatic system disorders) | 9 | 6
Anorexia (Metabolism and nutrition disorders) | 11 | 6
Anxiety (Psychiatric disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Blood bilirubin increased (Investigations) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Breast infection (Infections and infestations) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Chills (General disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 8 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Depression (Psychiatric disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 10 | 4
Dizziness (Nervous system disorders) | 3 | 3
Dry mouth (Gastrointestinal disorders) | 10 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 5
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Edema limbs (General disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 2 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 29 | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 4 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flu like symptoms (General disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 2
General disorders and administration site conditions - Other (General disorders) | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Gum infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 7 | 3
Hematuria (Renal and urinary disorders) | 0 | 1
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hot flashes (Vascular disorders) | 1 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 4
Investigations - Other (Investigations) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Movements involuntary (Nervous system disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 12 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 17 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Nervous system disorders - Other (Nervous system disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 5
Non-cardiac chest pain (General disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 3 | 1
Pain (General disorders) | 12 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 2
Peripheral motor neuropathy (Nervous system disorders) | 12 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 9
Platelet count decreased (Investigations) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Stomach pain (Gastrointestinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Tooth infection (Infections and infestations) | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 7 | 3
Urinary urgency (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Vascular disorders - Other (Vascular disorders) | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 7
Watering eyes (Eye disorders) | 3 | 1
Weight loss (Investigations) | 3 | 2
White blood cell decreased (Investigations) | 4 | 2

LIMITATIONS AND CAVEATS:
The study terminated early with cohort 2: TNBC not meeting target accrual of 45 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT01827787/Prot_SAP_000.pdf